CLINICAL TRIAL: NCT07178275
Title: The Effects of Qigong Exercises on Acute Anxiety, Mood, and Reaction Time Among Occupational Therapy Students: A Double-Blind, Crossover-Controlled Intervention Study
Brief Title: The Effects of Qigong Exercises on Acute Anxiety, Mood, and Reaction Time Among Occupational Therapy Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hulya YAMAN, Principal Investigator, Medipol University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4431
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: University Students

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized crossover study. Participants will be randomly assigned into two groups, defined as Group A and Group B. Following baseline assessments, Group A will receive a 60-minute Qigong intervention, while Group B will not receive any intervention and will remain in a resting condition. At the end of this first phase, outcome measures will be collected from both groups. After a one-day washout period to minimize potential carry-over effects, the groups will cross over. In the second phase, Group A will serve as the control with no intervention, while Group B will participate in the 60-minute Qigong session. Outcome measures will again be collected from both groups immediately following this phase.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong, Then Resting (Experimental): Participants first will receive a 60-minute Baduanjin Qigong session led by a licensed occupational therapist certified in Qigong. Qigong session will include gentle physical movements, controlled breathing, and meditative focus, performed in a quiet room under supervision. After a washout period of 1-day, participants will experience resting. In the resting time participants will undergo 60 minutes of passive rest in a quiet room. The use of phones, electronic devices, or any distracting materials will not be permitted.
  Interventions: Behavioral: Baduanjin Qigong; Behavioral: Passive Rest
- Resting, Then Qigong (Experimental): Participants first will undergo 60 minutes of passive rest in a quiet room. The use of phones, electronic devices, or any distracting materials will not be permitted. After a washout period of 1-day, participants will experience a 60-minute Baduanjin Qigong session led by a licensed occupational therapist certified in Qigong. The Qigong session will include gentle physical movements, controlled breathing, and meditative focus, performed in a quiet room under supervision.
  Interventions: Behavioral: Baduanjin Qigong; Behavioral: Passive Rest

INTERVENTIONS:
Behavioral: Baduanjin Qigong — A standardized 60-minute Baduanjin Qigong protocol (15 minutes of breathing-focused warm-up, eight movements each lasting 5 minutes, and 10 minutes of breathing-focused closing). The sessions will be conducted by a licensed occupational therapist certified in Qigong.
Behavioral: Passive Rest — Passive rest refers to a condition in which participants remain seated or lying quietly in a calm environment for a specified period of time, without engaging in any structured physical activity, therapeutic exercise, or cognitive tasks. During this period, external stimuli such as phone use, electronic devices, or reading materials are restricted in order to minimize distraction. The purpose of the passive rest condition is to provide a neutral control state that accounts for the passage of time and environmental factors, allowing valid comparison with the active intervention

SUMMARY:
The goal of this study is to examine the short-term effects of a single session of Baduanjin Qigong, a traditional mind-body exercise, on anxiety, mood, and reaction time in young adults studying occupational therapy. Baduanjin is a gentle form of Qigong that combines slow and rhythmic movements, breathing awareness, and mental focus. It has been practiced for centuries in China and has recently gained attention worldwide as a complementary therapy for improving mental, physical, and cognitive health.

University students are an important group to study because they often experience high levels of stress due to academic pressure, economic uncertainty, social expectations, and concerns about the future. These factors can increase vulnerability to problems such as anxiety, depression, attention difficulties, and sleep problems. While many studies have explored long-term non-drug interventions, there are still very few trials investigating immediate, short-term benefits of Qigong in young adult populations.

Previous research has shown that Baduanjin Qigong can reduce stress, anxiety, and depression, while also improving mood and physical health. For example, studies with college students have reported reductions in anxiety and depression, improvements in body mass index, lung function, and overall well-being after regular Baduanjin practice. Meta-analyses suggest that Baduanjin is especially effective in lowering stress compared to other traditional exercises. Some studies even found that just one 60-minute Qigong session can significantly reduce anxiety and improve mood, as measured by standard psychological tools. These findings suggest that Qigong can work not only as a long-term therapy but also as a rapid relief method in stressful situations.

In Turkey, most Qigong studies have focused on older adults or patient groups, showing benefits such as improved balance, reduced risk of falls, and better sleep quality. However, there are almost no experimental studies on the acute (short-term) psychological and cognitive effects of Qigong in young adults. This study aims to fill that gap.

What will happen in this study?

The study will recruit occupational therapy students.

Each participant will attend a single 60-minute Baduanjin session.

The design is double-blind, randomized, and crossover, which means that participants and evaluators will not know which condition they are assigned to, and each participant will experience both the Qigong session and a control condition on different days.

A short "wash-out" period will separate the sessions to ensure accurate results.

What will be measured?

Participants' anxiety, mood, and reaction time will be tested before and after the Qigong session.

Anxiety will be measured using the State-Trait Anxiety Inventory (STAI-Y1).

Mood will be measured using the Profile of Mood States (POMS).

Reaction time will be measured using a computerized test.

Why is this important?

This study will help us understand whether a single Qigong session can provide immediate psychological relief and improve mental focus for university students. If effective, Qigong could be considered a simple, low-cost, and accessible complementary practice to support student well-being in academic and daily life. The findings may also contribute to future health promotion programs targeting young adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 years
* Being an undergraduate occupational therapy student at Medipol University
* No history of chronic disease, psychiatric diagnosis, or condition preventing participation in physical exercise
* No prior regular participation in Qigong, yoga, or similar mind-body practices
* Voluntary participation and provision of informed consent

Exclusion Criteria:

* Use of antidepressant or psychotropic medication
* Acute pain, infection, or chronic cardiorespiratory disease
* Inability to complete computer-based visual reaction time testing

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
State Anxiety (STAI-Y1) | Both at the start and end of all interventions within one hour
  State anxiety (STAI-Y1) will be assessed using the State-Trait Anxiety Inventory, a validated self-report questionnaire. STAI-Y-1 scores range from 0 to 80 and higher scores are indicative of higher levels of state-anxiety

SECONDARY OUTCOMES:
Mood Profile (POMS) | Both at the start and end of all interventions within one hour
  Mood states will be measured using the Profile of Mood States (POMS), a standardized psychometric instrument. The Mood Scale is developed to assess short-term mood changes and consists of 65 words and 6 subscales. It is used to determine how participants feel before starting the test.
  Each individual rates the emotion/mood they experience on a Likert scale ranging from 1 ("not at all") to 5 ("extremely"). These 65 words correspond to six subscales: tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment.

OTHER OUTCOMES:
Reaction Time | Both at the start and end of all interventions within one hour
  Reaction time will be measured using a computer-based visual stimulus test assessing response latency in milliseconds. In the Go/No-go task, blue and red signals alternated as Go or No-go stimuli. Each was presented for 100 ms at 1,500-1,800 ms intervals, with 500 trials (30% Go) divided into five blocks. Participants pressed a button for Go and withheld responses for No-go.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim E, Lee JE, Sohn M. The Application of One-Hour Static Qigong Program to Decrease Needle Pain of Korean Adolescents With Type 1 Diabetes: A Randomized Crossover Design. J Evid Based Complementary Altern Med. 2017 Oct;22(4):897-901. doi: 10.1177/2156587217722473. Epub 2017 Aug 4. PMID 28776413
- [Background] Alkhatib A, Alshikh Ahmad H, Zhang C, Peng W, Li X. Impact of traditional Chinese Baduanjin exercise on menstrual health among international female students studying in China: a randomized controlled trial. Front Public Health. 2024 Feb 7;12:1259634. doi: 10.3389/fpubh.2024.1259634. eCollection 2024. PMID 38384881
- [Background] Luo X, Zhao M, Zhang Y, Zhang Y. Effects of baduanjin exercise on blood glucose, depression and anxiety among patients with type II diabetes and emotional disorders: A meta-analysis. Complement Ther Clin Pract. 2023 Feb;50:101702. doi: 10.1016/j.ctcp.2022.101702. Epub 2022 Nov 8. PMID 36423358
- [Background] Song, Y., Yang, Y., Dong, Y., & Li, S. (2021). Effects of aerobic exercise, traditional Chinese exercises and meditation on depressive symptoms of college students: A systematic review and network meta-analysis. Psychology, Health & Medicine, 27(6), 1321-1335.
- [Background] Rodrigues, D. F., Rosa, F. T., Lima, R. A., Oliveira, M. C., & Oliveira, D. V. (2021). Assessment of Qigong effects on anxiety of high school students: A randomized controlled trial. Complementary Therapies in Clinical Practice, 43, 101348. https://doi.org/10.1016/j.ctcp.2021.101348
- [Background] Wang X, Wu J, Ye M, Wang L, Zheng G. Effect of Baduanjin exercise on the cognitive function of middle-aged and older adults: A systematic review and meta-analysis. Complement Ther Med. 2021 Jun;59:102727. doi: 10.1016/j.ctim.2021.102727. Epub 2021 Apr 30. PMID 33933577
- [Background] Liu X, Li R, Cui J, Liu F, Smith L, Chen X, Zhang D. The Effects of Tai Chi and Qigong Exercise on Psychological Status in Adolescents: A Systematic Review and Meta-Analysis. Front Psychol. 2021 Nov 24;12:746975. doi: 10.3389/fpsyg.2021.746975. eCollection 2021. PMID 34899487

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT07178275/Prot_SAP_000.pdf